CLINICAL TRIAL: NCT07242677
Title: Post-market Observational Clinical Study With the Medical Device 'SPHEREPLAST' (SPHERE Study)
Brief Title: Post-market Observational Clinical Study With the Medical Device 'SPHEREPLAST'
Status: Not yet recruiting | Type: Observational
Sponsor: MT Ortho s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSMT-004
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Vertebra Compression Fracture; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, single-centre, single-arm post-market observational study evaluating the safety and clinical performance of the SPHEREPLAST medical device used in balloon kyphoplasty procedures for the treatment of traumatic and osteoporotic vertebral compression fractures (VCFs).

SPHEREPLAST is a titanium alloy (Ti6Al4V-ELI) trabecular sphere system designed to stabilise the vertebral body structure after balloon kyphoplasty, providing immediate mechanical stability and promoting bone ingrowth.

The study includes 40 adult patients who have been treated with SPHEREPLAST for thoracolumbar VCFs (A1, A3, OF2, OF3). Data will be collected retrospectively from medical records at four timepoints: pre-operative (baseline), within five days after surgery, at one month, and at one year post-surgery.

The primary endpoints are the changes in pain intensity (Numerical Rating Scale, NRS) and disability (Oswestry Disability Index, ODI) between baseline and 1-year follow-up. Secondary endpoints include radiographic outcomes (kyphotic angle, wedge angle, vertebral body height) and the incidence of adverse events related to the device or the procedure.

The aim of the study is to assess the real-world clinical efficacy and safety of SPHEREPLAST as an alternative to bone cement in kyphoplasty, with specific attention to pain control, functional recovery, and vertebral stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with SPHEREPLAST for post-traumatic thoracolumbar VCFs A1 and A3, osteoporotic OF2 and OF3;
* Complete availability of X-rays/MRI/CT scans;
* Painful vertebral fracture with bone oedema on MRI and at least NRS >4 units;
* At least 12 months of follow-up.

Exclusion Criteria:

* VCF associated with metastatic lesions and myeloma;
* Neurological impairment with compression of the spinal cord or nerves;
* General contraindications to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are men and women over the age of 18 treated with SPHEREPLAST for post-traumatic and osteoporotic thoracolumbar vertebral compression fracture
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
NRS (Numerical Rating Scale) | between baseline (pre-operative) and 1-year follow-up
ODI (Oswestry Disability Index) | between baseline (pre-operative) and 1-year follow-up

SECONDARY OUTCOMES:
adverse events (AEs), serious adverse events (SAEs) and adverse device events (ADEs) | postoperatively, at 1 month and at 1 year
NRS (Numerical Rating Scale) | baseline (pre-operative) and immediate post-operative and 1-month follow-ups
Kyphotic Angle (KA) | post-operative and 1-year follow-up
Wedge Angle (WA) | post-operative and 1-year follow-up
vertebral body height (VBH) | baseline, immediate post-operative and 1-year follow-up
  vertebral body height (VBH) in the anterior, middle and posterior projections

CONTACTS AND LOCATIONS:
Locations (1):
- G. Rodolico - San Marco University Hospital, Via S. Sofia, 78, Catania, CT, Italy